CLINICAL TRIAL: NCT05937711
Title: The Effect of Transcutaneous Posterior Tibial Nerve Stimulation on Pain and Quality of Life in Patients With Fibromyalgia: a Single-blind, Randomized Controlled Trial
Brief Title: The Effect of Transcutaneous Posterior Tibial Nerve Stimulation in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilker Fatih Sari (Other)
Responsible Party: Sponsor-Investigator, Ilker Fatih Sari, Assistant Professor, Giresun University
Organization: Giresun University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 90139838-000-E.61673
Record Dates: First submitted 2023-06-24; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
Keywords: Chronic pain; Electric stimulation therapy; Fibromyalgia; Quality of life; Small fiber neuropathy
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Small Fiber Neuropathy | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measures were assessed by investigators who were blinded to each patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTNS+Duloxetine (Experimental): Posterior tibial nerve stimulation (PTNS), twice weekly, 3-4 days apart + Duloxetine 30 mg 1X1 p.o PTNS was applied using two 50 mm × 50 mm electrode pads per extremity. The live pad was placed superior to and medial to the medial malleolus. The ground pad was placed 5-10 cm proximal to the live pad. The PTNS was applied using biphasic square waves with a frequency of 10 Hz and pulse duration of 200 μs. The amplitude was adjusted to the level that produced painless paresthesia in each patient according to their tolerance. PTNS was applied for 30 minutes
  Interventions: Other: Transcutaneous Posterior Tibial Nerve Stimulation + Duloxetine 30 MG; Drug: Duloxetine 30 MG
- Duloxetine (Active Comparator): Duloxetine 30 mg 1X1 p.o
  Interventions: Drug: Duloxetine 30 MG

INTERVENTIONS:
Other: Transcutaneous Posterior Tibial Nerve Stimulation + Duloxetine 30 MG — PTNS was applied using two 50 mm × 50 mm electrode pads per extremity. The live pad was placed superior to and medial to the medial malleolus. The ground pad was placed 5-10 cm proximal to the live pad. The PTNS was applied using biphasic square waves with a frequency of 10 Hz and pulse duration of 200 μs. The amplitude was adjusted to the level that produced painless paresthesia in each patient according to their tolerance. PTNS was applied for 30 minutes
  Duloxetine 30 mg p.o 1X1 (daily)
  Arms: PTNS+Duloxetine
Drug: Duloxetine 30 MG — Duloxetine 30 mg p.o 1X1 (daily)

SUMMARY:
This study aimed to investigate the effectiveness of posterior tibial nerve stimulation (PTNS) in reducing pain, improving quality of life, and decreasing disease severity in patients with fibromyalgia.

DETAILED DESCRIPTION:
This prospective, single-blind, randomized controlled trial included female patients newly diagnosed with fibromyalgia who had started duloxetine treatment (30 mg/day). Patients who met the inclusion criteria and agreed to participate in the study were randomized (1:1) into two groups. Group 1 (PTNS+duloxetine) underwent six sessions of posterior tibial nerve stimulation, twice weekly, 3-4 days apart, in addition to duloxetine (30 mg/day). Group 2 (duloxetine) received duloxetine only (30 mg/day). Randomization was performed manually, with assignments placed in opaque and sequentially numbered envelopes by off-site researchers who were not involved in patient care or follow-up. Outcome measures were assessed by two investigators who were blinded to each patient's group. The participants and nerve stimulators were not blinded to the group allocation. Patients were briefed to not disclose which group they were in during the assessment process.Patients in the study group received six sessions of posterior tibial nerve stimulation, twice weekly, 3-4 days apart, in addition to duloxetine; the controls received duloxetine only. The patients were evaluated three times (at baseline, 1st month, and 3rd month). Pain was evaluated using a numeric rating scale, the short-form McGill Pain Questionnaire, and quality of life with a 36-item Short-Form Health Survey (SF-36). Patient functional status and disease severity were evaluated using the fibromyalgia impact questionnaire (FIQ).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 65 years, newly diagnosed according to the American Rheumatology Association 2016 revised FMS diagnostic criteria
* Patients who come regularly to sessions for posterior tibial nerve stimulation.

Exclusion Criteria:

* History of fracture/musculoskeletal surgery in the last 3 years
* Inflammatory joint disease, or neurological disease/neurological deficit with examination
* Receiving medical treatment for polyneuropathy
* Contraindications to PNS (pacemaker, epilepsy, diminished skin sensation in the area to be applied).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since fibromyalgia is more common in women, female patients were included in the study.
Enrollment: 64 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Numeric Rating Scale (NRS) of pain score at week 4 and 12 | At baseline, 4th week and 12th week
  NRS was used to evaluate the patients' general pain at rest and during activity (during activities of daily living). Patients were asked to rate their pain from 0 to 10, with 0 indicating no pain and 10 indicating the most severe pain
Change from baseline in Short-Form McGill Pain Questionnaire at week 4 and 12 | At baseline, 4th week and 12th week
  This questionnaire was used to assess the patients' pain. This questionnaire consisted of 15 descriptive words that evaluated the sensory (11) and affective (4) dimensions of pain. Pain intensity was evaluated as follows: 0=none, 1=mild, 2=moderate, and 3=severe. Three pain scores were obtained: sensory, affective, and total (both sensory and affective). The total present pain intensity index was evaluated using a 6-point Likert rating scale. (0 = no pain, 1 = mild, 2 = discomforting, 3 = distressing, 4 = horrible, and 5 = excruciating)

SECONDARY OUTCOMES:
Change from baseline in Fibromyalgia Impact Questionaire at week 4 and 12 | At baseline, 4th week and 12th week
  This questionnaire consists of 20 questions evaluating physical function, job status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being of patients with fibromyalgia. It was scored between 0 and 100. High scores indicate high disease severity and low functional status.
Change from baseline in The 36-item Short-Form Health Survey at week 4 and 12 | At baseline, 4th week and 12th week
  This scale is commonly used to evaluate the quality of life. It consists of eight subscales (physical function, physical role limitation, pain, general health, vitality, social function, social role limitation, and mental health) and a total of 36 items. Each subscale was scored between 0 and 100, with 100 points indicating the best health condition and 0 points indicating the worst health condition

CONTACTS AND LOCATIONS:
Overall Officials: İlker Fatih Sarı, Principal Investigator — Giresun University Faculty of Medicine, The Department of Physical Medicine and Rehabilitation
Locations (2):
- Turkey (Türkiye) (2):
  - Giresun University Faculty of Medicine, Giresun
  - Ondokuz Mayıs University Faculty of Medicine, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295
- [Background] Cheng CW, Wong CS, Hui GK, Chung EK, Wong SH. Fibromyalgia: is it a neuropathic pain? Pain Manag. 2018 Sep 1;8(5):377-388. doi: 10.2217/pmt-2018-0024. Epub 2018 Sep 13. PMID 30212264
- [Background] Uceyler N, Zeller D, Kahn AK, Kewenig S, Kittel-Schneider S, Schmid A, Casanova-Molla J, Reiners K, Sommer C. Small fibre pathology in patients with fibromyalgia syndrome. Brain. 2013 Jun;136(Pt 6):1857-67. doi: 10.1093/brain/awt053. Epub 2013 Mar 9. PMID 23474848
- [Background] Lin T, Gargya A, Singh H, Sivanesan E, Gulati A. Mechanism of Peripheral Nerve Stimulation in Chronic Pain. Pain Med. 2020 Aug 1;21(Suppl 1):S6-S12. doi: 10.1093/pm/pnaa164. PMID 32804230
- [Background] Slavin KV. Peripheral nerve stimulation for neuropathic pain. Neurotherapeutics. 2008 Jan;5(1):100-6. doi: 10.1016/j.nurt.2007.11.005. PMID 18164488
- [Background] Oaklander AL, Herzog ZD, Downs HM, Klein MM. Objective evidence that small-fiber polyneuropathy underlies some illnesses currently labeled as fibromyalgia. Pain. 2013 Nov;154(11):2310-2316. doi: 10.1016/j.pain.2013.06.001. Epub 2013 Jun 5. PMID 23748113
- [Background] Dabby R, Sadeh M, Goldberg I, Finkelshtein V. Electrical stimulation of the posterior tibial nerve reduces neuropathic pain in patients with polyneuropathy. J Pain Res. 2017 Nov 29;10:2717-2723. doi: 10.2147/JPR.S137420. eCollection 2017. PMID 29238215
- [Background] Thimineur M, De Ridder D. C2 area neurostimulation: a surgical treatment for fibromyalgia. Pain Med. 2007 Nov-Dec;8(8):639-46. doi: 10.1111/j.1526-4637.2007.00365.x. PMID 18028042
- [Derived] Sari IF, Ilhanli I, Mizrak T, Kulakli F, Kasap Z. The Effect of Transcutaneous Posterior Tibial Nerve Stimulation on Pain and Quality of Life in Patients with Fibromyalgia: A Single-Blind, Randomized Controlled Trial. J Clin Med. 2023 Jul 29;12(15):4989. doi: 10.3390/jcm12154989. PMID 37568391